CLINICAL TRIAL: NCT01476176
Title: A Pivotal Pharmacokinetic Study Investigating the Extent of Absorptions of Paracetamol and Caffeine for Two Different Paracetomol Formulations Containing Caffeine
Brief Title: A Pharmacokinetic Study of an Experimental Paracetamol Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: A2260665
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-06

CONDITIONS: Headache, Tension-Type
Keywords: Bioequivalence; Pharmacokinetics; Healthy volunteers; paracetamol; caffeine
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental paracetamol formulation (Experimental): experimental formulation
  Interventions: Drug: Experimental paracetamol
- paracetamol marketed formulation (Active Comparator): Paracetamol marketed formulation
  Interventions: Drug: Paracetamol marketed formulation

INTERVENTIONS:
Drug: Experimental paracetamol — experimental paracetamol with caffeine
  Arms: Experimental paracetamol formulation
Drug: Paracetamol marketed formulation — marketed formulation containing caffeine
  Arms: paracetamol marketed formulation

SUMMARY:
This PK study is designed to show bioequivalence between the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
PK variables (AUC 0-10hrs, AUC 0-inf, and Cmax) to determine bioequivalence | 10 hours

SECONDARY OUTCOMES:
PK variables to compare speed of absorption (AUC 0-30min, AUC 0-60min, Tmax) | 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- MDS Pharma Services ARIZONA, Phoenix, Arizona, United States